CLINICAL TRIAL: NCT05023200
Title: The Personalised Antibiotic Duration for Cellulitis (PAD-C) Cohort Study
Brief Title: The Personalised Antibiotic Duration for Cellulitis (PAD-C) Study
Acronym: PAD-C
Status: Completed | Type: Observational
Sponsor: University of Sussex (Other)
Responsible Party: Principal Investigator, Elizabeth Cross, Chief Investigator, University of Sussex
Other Study IDs: 081 CRO / 295690; NIHR300952 (Other: NIHR Doctoral Fellowship); 295690 (Other Grant/Funding Number: IRAS)
Record Dates: First submitted 2021-08-12; First posted 2021-08-26 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Cellulitis; Cellulitis of Leg; Antibiotic Duration
Keywords: Cellulitis; Antibiotics; Treatment duration; Treatment length
MeSH Terms: conditions — Cellulitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Population: Adults (age ≥18 years) identified by their treating clinician as having lower limb cellulitis that requires intravenous or oral antibiotic treatment either from the hospital or another service based outside of the hospital, which will conduct ongoing follow-up regardless of location.

SUMMARY:
Cellulitis is an increasingly common and unpleasant bacterial infection of the skin, usually affecting the legs. Patients experience pain and swelling, loss of mobility, fever, and chills. Patients may be left with chronic skin damage and 1 in 5 experience recurrences.

Cellulitis is treated with antibiotics, but it is unclear as to how long treatment should be for. As a result, many patients get much longer antibiotic treatment than needed. This exposes patients to the risks of taking unnecessary antibiotics.

This study aims to find out what features of individual patients predict a good, sustained recovery from cellulitis. These may include medical conditions and clinical response to the first few days of antibiotic treatment, such as changes in skin temperature.

Patients who are being treated in hospital for cellulitis will be invited to take part. Information will be collected about patients who will be followed up for 3-6 months. Devices for measuring skin temperature will also be compared to see which one works best. This information will be used to help develop a set of rules that doctors can use to guide the length of antibiotic treatment. This should ensure that future patients receive the amount of antibiotics needed and no more.

DETAILED DESCRIPTION:
This study is a single centre prospective cohort study of patients with cellulitis of the lower limb. The primary objective of this study is to understand what features of individual patients predict a sustained recovery from cellulitis. This information will be used to test and refine a previously developed risk score that predicts clinical outcomes of patients with cellulitis.

Secondary objectives include investigating whether early response to antibiotic treatment (e.g. reduction in skin temperature and patient-reported symptoms) improves the predictive ability of the risk score. The study design also includes a nested technology comparison of temperature measurement devices to identify the best device for measuring affected skin temperature change in patients with cellulitis.

Clinical response will be measured for up to four days from starting antibiotic treatment. This includes the change in temperature and area of affected skin, physiological observations, blood test results (e.g. C-reactive protein) and patient-reported pain and swelling scores. Patients will be followed up at 28 and 90 days (+/- 180 days for those recruited in the first year) to assess recovery, recurrence, cellulitis-related mortality, quality of life, and return to normal activities.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years) identified by their treating clinician as having lower limb cellulitis that requires IV or oral antibiotic treatment either from the hospital or another service based outside of the hospital, which will conduct ongoing follow-up regardless of location.

Exclusion Criteria:

Patients:

* who have already received 3 or more calendar days of antibiotics from the hospital for cellulitis.
* receiving antibiotic therapy for another indication that is anticipated to continue for longer than the antibiotic treatment for cellulitis and that, in the judgement of the investigator, would impact the study assessments.
* for whom a surgical procedure to treat their cellulitis is planned (i.e. debridement of suspected necrotising skin / soft tissue infection).
* who, in the judgement of the investigator, do not have a clear diagnosis of cellulitis (to enable the exclusion of infections, such as severe/deep diabetic foot infection, which may be loosely labelled as cellulitis, but treated with different guideline antibiotic agents and durations).
* lack capacity to give informed consent to participate.
* are receiving end-of-life care.
* are already involved in a CTIMP of relevance to the treatment of their cellulitis.
* are unlikely, in the opinion of the investigator, to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital-based or services delivering antibiotic treatment and ongoing follow-up regardless of location.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
Sustained recovery | 90 days
  No initiation of new antibiotic treatment for cellulitis at the same site through to 90 days

SECONDARY OUTCOMES:
Recovery at 28 days | 28 +/- 3 days
  The absence of warmth and tenderness at the site, with improvement in swelling and acute colour change, that did not require new antibiotic treatment
Patient-reported time to resolution of cellulitis symptoms | 28 +/- 3 days
  Patient-reported time to resolution of cellulitis and symptoms of pain and swelling, using a numeric and verbal marked scale (1 to 10, higher score indicates higher severity of symptom)
Change in quality of life | Baseline, 90 days (+/- 180 days for a subset recruited within the first year)
  Change in quality of life assessed using the Medical Outcomes Study Short Form 12-Item Health Survey (SF-12) compared to baseline
Time to return to work / normal activities | Baseline, 28 days, 90 days (+/- 180 days for a subset recruited within the first year)
  Patient-reported date at which they returned to work / normal activities
Cellulitis-related readmission | 90 days (+/- 180 days for a subset recruited within the first year)
  New hospital admissions/reattendance containing a cellulitis diagnostic code
Cellulitis-related mortality | 90 days (+/- 180 days for a subset recruited within the first year)
  Death within 90 (+/- 180) days of initial admission/attendance
Antibiotic usage and antibiotic-related adverse events | Through study completion, an average of 180 days
  Route and duration of antibiotic therapy, adverse events from patient-report, medical and laboratory records

OTHER OUTCOMES:
Repeatability coefficient | Measurements taken at 0 to 3 days
  Repeatability of the measurements taken by the temperature measurement devices
Limits of agreement | Measurements taken at 0 to 3 days
  Estimate of agreement between the temperature measurement devices quantified by estimating the limits of agreement

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth LA Cross, Principal Investigator — University of Sussex
Locations (1):
- University Hospitals Sussex NHS Foundation Trust, Brighton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised study data is intended to be made available via an open access research database.